CLINICAL TRIAL: NCT00442754
Title: Vaccination With Autologous Dendritic Cells Pulsed With Allogeneic Tumour Lysate (MelCancerVac) for the Treatment of Patients With Advanced or Metastatic Non-Small Cell Lung Cancer. A Phase II Study
Brief Title: Dendritic Cells in Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Dina rosenberg asmussen, Dandrit biotech
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dendric cells in lungcancer
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2009-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: dendritic cell; tumor vaccine; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Allogeneic Tumour Lysate (MelCancerVac) — subcutaneaus, /once weekly /4 wks then /4 weekly

SUMMARY:
Vaccination with autologous dendritic cells pulsed with allogeneic melanoma cell lysate (MelCancerVac) in combination with the Cox-2 inhibitor of celecoxib for the treatment of patients with advanced or metastatic non-small cell lung cancer (NSCLC). Adjuvant Aldara cream will be used as adjuvant for induction of inflammation at the injection site, and the lymphocyte growth factor of interleukin-2 (IL-2) will be given as s.c. injection. The treatment aims at boosting the patient's specific immune system against the cancer cells.

DETAILED DESCRIPTION:
Vaccination with autologous dendritic cells pulsed with allogeneic melanoma cell lysate (MelCancerVac) in combination with the Cox-2 inhibitor of celecoxib for the treatment of patients with advanced or metastatic non-small cell lung cancer (NSCLC). Adjuvant Aldara cream will be used as adjuvant for induction of inflammation at the injection site, and the lymphocyte growth factor of interleukin-2 (IL-2) will be given as s.c. injection. The treatment aims at boosting the patient's specific immune system against the cancer cells.

Patients with disseminated, inoperable NSCLC after chemotherapy and patients not wanting chemotherapy for which no other systemic treatments can be offered.

Primary objective: to measure the antigen specific immunological reaction between vaccine antigens and the patients' immune system in vivo and in vitro.

Secondary objectives: to estimate the patients' survival time, to estimate response according to RECIST criteria, and to estimate the patients' quality of life during the study period.

The study is designed as an open, phase II, clinical study and will be carried out in accordance with the present protocol, ICH/GCP Guidelines and national, regulatory requirements.

The first patient is expected to be included towards the end of 2006. Inclusion period will continue for 2 years. Follow-up will continue for approx. 6 months prior to reporting.

Fifty patients are planned for inclusion. In case none of the first fourteen (14) evaluable patients will respond, the inclusion and the study will be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Primary objective: to measure the antigen specific immunological reaction between vaccine antigens and the patients' immune system in vivo and in vitro. | 3 years

SECONDARY OUTCOMES:
Secondary objectives: to estimate the patients' survival time, to estimate response according to RECIST criteria, and to estimate the patients' quality of life during the study period. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: anders mellemgaard, MD PhD, Principal Investigator — Dept of Oncology, herlev university hospital
Locations (1):
- Herlev University Hospital, Copenhagen, Denmark